CLINICAL TRIAL: NCT00768131
Title: A Randomized Phase II Trial to Assess the Predictive Value of Increased EGFR Copy Number by FISH in Patients With Advanced / Metastatic NSCLC Treated With Cetuximab and Carboplatin / Paclitaxel
Brief Title: A Study to Determine Whether EGFR Status by FISH Can Predict Results in Non Small Cell Lung Cancer (NSCLC) Patients Treated With Cetuximab, Carboplatin and Paclitaxel
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CA225-322
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Lung Neoplasms; Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A1 FISH (+) (Experimental)
  Interventions: Drug: Cetuximab; Drug: Paclitaxel; Drug: Carboplatin
- B1 FISH (+) (Active Comparator)
  Interventions: Drug: Paclitaxel; Drug: Carboplatin
- A2 FISH (-) (Experimental)
  Interventions: Drug: Cetuximab; Drug: Paclitaxel; Drug: Carboplatin
- B2 FISH (-) (Active Comparator)
  Interventions: Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Cetuximab — Vial, Intravenous, 400 mg/m² week 1 then 250 mg/m², Weekly, Until PD/Toxicity/Pt-PI Decision
  Other Names: Erbitux; BMS-564717
  Arms: A1 FISH (+); A2 FISH (-)
Drug: Paclitaxel — Vial, Intravenous, 225 mg/m2, Every 3 weeks, 6 cycles maximum
Drug: Carboplatin — Vial, Intravenous, AUC = 6.0, Every 3 weeks, 6 cycles maximum

SUMMARY:
The purpose of this study is to determine if EGFR status (positive or negative) by FISH can predict response to cetuximab therapy in NSCLC patients treated with carboplatin and paclitaxel

ELIGIBILITY:
Inclusion Criteria:

* Subjects who present with Stage IV, Stage IIIB NSCLC or recurrent disease following radiation therapy or surgical resection
* No prior chemotherapy or anti-EGFR targeted therapy
* Sufficient tumor material for FISH testing
* Measurable disease (RECIST)
* ECOG performance status 0 or 1

Exclusion Criteria:

* Symptomatic or uncontrolled CNS metastases
* Inadequate hematologic function defined as ANC < 1,500/mm3, platelet count < 100,000/mm3, or a hemoglobin level < 9 g/dl
* Inadequate hepatic function defined as total bilirubin > 1.25 x ULN, AST level > 1.5 x ULN, or alkaline phosphatase > 5.0 x ULN
* Inadequate renal function defined by a serum creatinine level > 1.5 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) will be compared for FISH positive subjects (subset) receiving paclitaxel / carboplatin +/- cetuximab | Every 6 weeks

SECONDARY OUTCOMES:
Tumor response | Every 6 weeks
Disease control | Every 6 weeks
Overall survival (OS) | Every 4 months after subject off-treatment until 1 year after LPLT
Duration of Response | Every 6 weeks
Safety & exploratory biomarker analysis | Every 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- United States (14):
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Long Beach, California
  - Local Institution, Boynton Beach, Florida
  - Local Institution, Chicago, Illinois
  - Local Institution, Skokie, Illinois
  - Local Institution, Wichita, Kansas
  - Local Institution, Louisville, Kentucky
  - Local Institution, Mount Sterling, Kentucky
  - Local Institution, Annapolis, Maryland
  - Local Institution, Kalamazoo, Michigan
  - Local Institution, Staten Island, New York
  - Local Institution, Winston-Salem, North Carolina
  - Local Institution, Portland, Oregon
  - Local Institution, Austin, Texas

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx